CLINICAL TRIAL: NCT06374446
Title: Investigation of the Effect of Virtual Reality on Fatigue, Functional Capacity and Respiratory Function in Patients With Long Covid-19
Brief Title: Effect of Virtual Reality in Patients With Long Covid-19
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-172
Record Dates: First submitted 2024-01-25; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Classical Treatment (Experimental): Upper and lower extremity exercises + breathing exercises
  Interventions: Other: Classical Treatment
- Virtual Reality Combined with Classical Treatment (Experimental): Upper and lower extremity exercises + breathing exercises+virtual reality
  Interventions: Other: Virtual Reality Combined with Classical Treatment
- Virtual Reality Group (Experimental): Virtual reality
  Interventions: Other: Virtual Reality
- Control Group (Experimental): A brochure with home program explaining the importance of exercise will be given
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Classical Treatment — This group in our study exercises 2 days a week, 2 repetitions a day, 3 sets of 15 repetitions for 6 weeks. Upper and lower extremity exercises are available, including shoulder flexion and abduction, hip and knee exercises. Active breathing cycle is used as breathing exercises. Active respiratory cycle; Includes breathing control, thoracic expansion exercises and huffing. These are done for 6 weeks, along with upper and lower extremity exercises. All evaluations are made at the beginning and end of the groups.
  Arms: Classical Treatment
Other: Virtual Reality Combined with Classical Treatment — This group in our study exercises 2 days a week, 2 repetitions a day, 3 sets of 15 repetitions for 6 weeks. Upper and lower extremity exercises are available, including shoulder flexion and abduction, hip and knee exercises. Active breathing cycle is used as breathing exercises. Active respiratory cycle; Includes breathing control, thoracic expansion exercises and huffing. These are done for 6 weeks, along with upper and lower extremity exercises. In addition, individuals can take a 30-minute walk in the forest, do yoga, etc. with virtual reality glasses. Videos for relaxation will be shown. All evaluations will be made at the beginning and end of the groups.
  Arms: Virtual Reality Combined with Classical Treatment
Other: Virtual Reality — Individuals in this group are given 30-minute walks in the forest, yoga, etc. with virtual reality glasses, 2 days a week, 2 times a day for 6 weeks. Videos for relaxation will be shown. All evaluations will be made at the beginning and end of the groups.
  Arms: Virtual Reality Group
Other: Control Group — This group will be given a handbook explaining the importance of exercise in individuals with long-term symptoms after Covid.
  Arms: Control Group

SUMMARY:
SARS-CoV-2 was first detected in Wuhan, Hubei Province, China, in late 2019. It is a highly contagious virus that has been reported to occur in humans and is said to cause pneumonia.

Covid-19 infection is transmitted through droplets during coughing and sneezing and through contact with the mouth, nose or eyes after contaminated hands. The most obvious symptoms of Covid-19 symptoms include cough, dyspnea and fever. Covid-19, which can also be seen asymptomatic, is in intensive care it may be severe enough to require hospitalization, cause multiple organ failure and even death it could be. Musculoskeletal symptoms such as fatigue, myalgia, and arthralgia are common with Covid-19 are the symptoms. The first case in Turkey was reported on March 11, 2020.

Long-term Covid or Chronic Post Covid Syndrome are multi-system syndromes that last more than 12 weeks and physical, cognitive, psychological, social and occupational domains. The most commonly reported long covid symptoms are; fatigue, shortness of breath, cough, joint pain, chest pain.

Virtual reality application provides its users with content created using computer technology. In a virtual environment with a high perception of reality, the aim is to enable mirror neuron activation, enabling the individual to interact with virtual objects and events with three-dimensional movements and to create the perception of doing all these in the real world.

Virtual reality for training, treatment, rehabilitation, analysis and testing purposes in healthcare can be used. It is possible to use virtual reality for different purposes, for treatment and rehabilitation. With virtual reality applications in treatment and rehabilitation processes It was stated that patient motivation will increase and patient fear and anxiety will decrease.

No study was found in the literature investigating the effect of virtual reality application on fatigue, functional capacity and respiratory function in long-term Covid-19 patients. The purpose of this study; To investigate the effect of virtual reality application on fatigue, functional level and respiratory function in long-term Covid-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 - 65
* Having been diagnosed with Covid-19
* At least 12 weeks have passed since the diagnosis of Covid-19 and the symptoms continue
* To be cooperative

Exclusion Criteria:

* Having been KOAH
* People with severe visual and cognitive impairment
* Having a neuromuscular disease
* Having a cardiac or pulmonary surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 6 weeks
  It will be evaluated with the Visual Analog Scale. It will be used to objectively determine the degree of pain at rest and during activity. Visual Analogue Scale is a 10 cm line drawn in the horizontal plane on a white sheet of paper. The words "no pain" are on the left end and "the most severe pain you have ever encountered in your life" are on the right. It was explained to the patient that the severity of pain increased from left to right, and he was asked to mark the severity of his own pain separately on this line at rest and during movement. There will be 2 different evaluations as Visual Analogue Scale-Rest and Visual Analogue ScaleActivity. Evaluations will be measured at the start of treatment and at the end of the study.
Kinesiophobia | 6 weeks
  Kinesiophobia means fear of movement. Tampa Kinesiophobia Scale consists of 17 items. It determines the impact of injury and fear on the inability to perform movements in daily life and activities. In questions, the patient ticks the box for the answer he finds appropriate. The score for each question is determined by the answer. There is a score range of 1-4. The overall score is in the range of 17-68. The total score is calculated after reversing items 4, 8, 12 and 16. The higher the total score, the higher the level of kinesiophobia.
Evaluation of Respiratory Function | 6 weeks
  It is performed with a respiratory function test. It is performed with a spirometer device according to the American Thoracic Society and European Respiratory Society criteria; forced vital capacity (FVC), forced expiratory volume (FEV1), forced expiratory volume/ forced vital capacity (FEV1/FVC), 20 peak expiratory flow (PEF) and forced expiratory flow 25-75% (FEF25-75%) values are recorded.
Shuttle Walking Test | 6 weeks
  This test is an exercise test in which you walk for 12 minutes at increasing speed between two cones 10 m apart, with each 10-meter journey between the two cones counting as one shuttle. Testing is continued until the patient is unable to continue testing due to shortness of breath, the heart rate reaches 85% of the maximum expected heart rate, or the test is completed for 12 minutes. What is actually measured in this test is the distance walked. It is calculated based on the number of sit-ups completed. In healthy people, a walking distance of 824 m can be reached between the ages of 40-49, 788 m between the ages of 50-59, 699 m between the ages of 60-69, and 633 m for people aged 70 and over. .
Endurance Shuttle Walking Test | 6 weeks
  Endurance Shuttle Walking Test In this test, you walk at a constant speed between cones 10 m apart. The selected speed is 85% of the person's maximum capacity measured in the shuttle walking test at increasing speed. Therefore, before this test, the patient must undergo a shuttle walking test at an increased speed. The test is terminated in 20 minutes. It is a test developed to determine submaximal exercise capacity in daily living activities. It is aimed to eliminate individual differences by directing the walking speed externally with audible signals. In this test, walking time, heart rate, oxygen saturation and dyspnea level are measured.
Sit and Reach Test | 6 weeks
  It was used to measure hamstrings flexibility. The test was performed by measuring the distance from the hands to the tip of the toes while the patient was in a long sitting position in bed, without bending his knees. His last destination was recorded. If the hands did not touch the feet, the values were recorded as negative, if they passed the feet, the values were recorded as positive.
Peripheral Muscle Strength | 6 weeks
  It will be evaluated with a hand dynamometer and myometer. Hand grip strength is a simple measurement method used to measure upper extremity function. Measurement of hand grip strength is used in many studies in the field of pulmonary rehabilitation because it is an easy and useful method. There are different types of dynamometers. However, the Jamar hand dynamometer, which has high validity and reliability, is recommended by the American Association of Hand Therapists, and is considered the gold standard, is used in the studies. Elbow and shoulder flexors, shoulder abduction and knee extension will be measured with a myometer. Tests will begin to be administered after detailed information about how the test is performed and a trial has been carried out once. The measurements will be repeated 3 times and the arithmetic average will be accepted as the value taken by the device and will be recorded on the patient follow-up forms.
The Nottingham Health Profile | 6 weeks
  The Nottingham Health Profile will be used in our quality of life assessment. In the questionnaire consisting of 38 items, 6 different parameters related to health status are evaluated. These parameters are physical activity (8 items), emotional reactions (9 items), energy (3 items), social isolation (5 items), pain (8 items), and sleep (5 items). Each subparameter is scored between 0-100. A high score indicates worsening health. The total score is obtained by summing all sub-parameter scores.
Dyspnea | 6 weeks
  Individuals is dyspnea level will be measured using the Modified Medical Research Council (MMRC) Dyspnea Scale. The scale, which was created considering different physical activities that cause the feeling of dyspnea, has five items and the scoring is between 0-4 points. 0: no shortness of breath except during strenuous exercise, 1: shortness of breath when rushing on level ground or going up a slight incline, 2: walking slower than people of the same age due to shortness of breath or having to stop for breath when walking at their own pace on the level; 3: Pauses for breath after walking ∼100 m or after a few minutes at the level, 4: Too out of breath to leave the house or out of breath when dressing or undressing
Energy Consumption | 6 weeks
  ActiGraph wGT3X-BT device is used for objective measurement of physical activity. It is a device worn on various parts of the body, mostly on the thigh, ankle, waist and wrist, that records physical movement associated with daily living activities and sleep. Data regarding the number of steps and time spent in different physical activity intensities are obtained with the device. It is requested that the attached devices should not be removed for 7 days, except for swimming, bathing and water-requiring situations. The epoch length of the device should be set to 1, 5, 15, 30 or 60 seconds. It must be worn at least 4 days a week, including one on the weekend, and at least 10 hours a day. ActiGraph energy expenditure is estimated by calculating the vector size. Predictive equations have been developed to convert these numbers into units of energy expenditure. Energy consumption is calculated in METs or kilocalories. It is considered the gold standard in terms of energy consumption.
Posture Analysis | 6 weeks
  Corbin et al.'s form will be used when performing posture evaluation on individuals. This form is based on scoring postural disorders observed from the lateral and posterior according to their severity (0: none, 1: mild, 2: moderate, 3: severe). It also allows classifying the individual's postural status according to the total scores obtained. Observations are analyzed from posterior and lateral regions
Covid-19 Yorkshire Performance | 6 weeks
  C19-YRS consists of 22 items, with each item rated on an 11-point numerical rating performance from 0 to 10. The C19-YRS is divided into four subscales (total score range for each subscale): symbol gender score (0-100), functional disability score (0-50), supplementary score (0-60), and general health (0-10). )
FACIT Fatigue Scale | 6 weeks
  There are 13 questions in this dimension, detailed by Tennant et al., for the objective assessment of fatigue. This test, which has 5 options such as not at all, very little, a little, a lot and a lot, should be taken into consideration for the last week when filling out. The feeling of fatigue and burnout that the person encounters in his daily life and activities will be questioned

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Buran Çırak, Prof., Principal Investigator — Istinye University

IPD SHARING:
Plan to Share IPD: No